CLINICAL TRIAL: NCT05358470
Title: Effects of a Exercise Therapy Program Based on Sports Towards People With Acquired Brain Injury: a Randomized Controlled Trial
Brief Title: Exercise Therapy Program on Acquired Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade da Coruña (Other)
Responsible Party: Principal Investigator, Beatriz Rodríguez-Romero, Lecturer at Department of Physiotherapy, Medicine and Biomedical Sciences. Universidade da Coruña, Universidade da Coruña
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: Exercise-acquired brain injury
Record Dates: First submitted 2022-03-21; First posted 2022-05-03 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Acquired Brain Injury
Keywords: Exercise therapy; Physical Therapy; Exercise; Sports for persons with disabilities
MeSH Terms: conditions — Brain Injuries; Motor Activity | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise therapy and adapted physical activity-based intervention (Experimental): The intervention in the experimental group (EG) consists of a exercise therapy and adapted physical activity program based on racket sports. The immediate EG will receive sixteen, twice a week, one-hour sessions of group-based, racket sports specific fundamental movement skills training. All sessions will be guided and supervised by a physiotherapist and delivered in groups of 5 participants to promote exchange and conviviality and to optimize the rates of participation and compliance.
  Interventions: Other: Exercise therapy and adapted physical activity-based program
- Usual care (No Intervention): Participants in the CG receive conventional management with general physical activity recommendation.

INTERVENTIONS:
Other: Exercise therapy and adapted physical activity-based program — Exercise therapy and adapted physical activity program based on racket sports
  Arms: Exercise therapy and adapted physical activity-based intervention

SUMMARY:
In this study, the physical and psychosocial effects of a exercise therapy and adapted physical activity program based on racket sports for ambulant people with acquired brain injury will be investigated.

DETAILED DESCRIPTION:
The proposed protocol study is a two-arm, randomized, assessor-blinded trial with two parallel groups.

The study population consists of ambulant people aged more than 18 years with a confirmed diagnosis of acquire brain injury at subacute or chronic stages. Participants who agree to participate in the study will be assigned to experimental group (EG) (exercise therapy and adapted physical activity program) or control group (CG) (usual care) after being screened and randomized according to the inclusion criteria.

A physiotherapist will perform the evaluation process, including physical performance and biopsychosocial aspects. Information on functioning and disability will be collected through the ICF components, including Contextual Factors such as "Personal" and "Environmental", and Functioning domains such as "Body Functions and Structures" (b-components), "Activities & Participation" (d-components) as well as "Quality of Life components" . The main outcome measures of the study are: (i)"health-related quality of life" through the questionnaire Short Form 36; (ii) "functional capacity", attending to aspects of mobility and endurance on walking which will be measured through two tests: the 6 Minutes Walk Test and the 10 Meter Walk Test; (iii) motor control of the upper limb, through the Fugl-Meyer Upper Extremity test; (iv) "mobility" which will be measured with Timed Up and Go; (v) and "balance", through the Balance Berg Scale. As secondary outcome measures of the study, the level of physical activity through the Global Physical Activity Questionnaire will be measured. Moreover, demographic and anthropometric characteristics will be also considered.

Outcome measures will be assessed at baseline (T1) and immediately after 8 weeks of program (T2),

Participants in EG a progressive program based on a therapeutic exercise and adapted physical activity program based on racket sports, will be practiced for 60 minutes a day, 2 days a week for 8 weeks. In CG, participants will receive conventional management with general physical activity recommendation. The intervention will be guided and supervised by a physiotherapist and delivered in groups of 5 participants.

Randomization process (sequence generation, allocation concealment, and implementation) will be conducted by three different researchers from the team. After signing the informed consent and undergoing initial assessment, participants will be allocated to the experimental group (EG) or the control group (CG). It will be made using a computer-generated number sequence, with a 1:1 allocation ratio, without stratification.

The assessments (T1, T2) will be completed by two physiotherapists specifically trained to carry out the outcomes evaluations who will be blinded to group allocation during the entire study period.

The sample size is estimated to obtain statistically significant improvements through the two primary outcomes: (i) health-related quality of life (Physical Component Summary) and (ii) functional capacity (6-minute walk).

(i)The threshold for detecting changes in health-related quality of life is approximately 5 points (Norman et al. 2003). To detect this difference with a standard deviation (SD) of ±5 points between the groups with a 95% confidence interval and a statistical power of 80% in a two-side approach, it would be needed 16 participants. Considering that it could have 15% losses, the final sample size would be 18 subjects in each group.

(ii) On the other hand, since there are no published data on the 6-minute walk test in adults with ABI, it is considered the clinical difference to be significant in healthy adults (standard deviation of ±44). To detect the difference between groups with a confidence interval of 95% and a statistical power of 80%, the sample should be composed of 12 persons by group. Considering a 15% losses, the final sample size would be 14 participants in each group.

In addition, based on previous studies that carried out a similar intervention in persons with adquired brian injury, the total sample should ranged between 30-35 participants.

Both ethics approval and administrative site approvals have been granted by the local ethics committee (Ethics Committee for Clinical Investigation of Madrid, Spain). Full written informed consent will be obtained from all participants indicating voluntary participation in the study. All informed consent data will be collected and stored by the main researcher. This clinical trial has been performed in accordance with the Helsinki Declaration. Participants' personal data will be de-identified (they will be allocated a identification code generated by a random number sequence, which will be used to deidentify participant information). No data that could identify the participants will be published.

ELIGIBILITY:
Inclusion Criteria:

* Persons with a medical diagnosis of acquired brain injury in subacute or chronic stages.
* To be aged >18 years at study entry
* To have an independent gait without the need of technical aids: a score of 3, 4 or 5 from the Functional Ambulation Categories (FAC) walking test.
* Be able to understand simple instructions from the program protocols as well as perform baseline and post-intervention assessments.

Exclusion Criteria:

* Not have a completed and signed informed consent form.
* Non-attendance and/or non-collaboration to 70% of the program sessions.
* To have medical co-morbidities that contraindicate physical exercise safely (e.g. cardiac or respiratory instability, uncontrolled seizures)
* Non-collaboration during the pre- and post-tests of the program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Functional capacity: 10 Meter Walk Test | Baseline, Change from Baseline at 8th week
  - 10 Meter Walk Test: The 10MWT is a performance measure used to assess walking speed in meters per second over a short distance. It can be employed to determine functional mobility, gait, and vestibular function.
Motor control of the upper limb test: Fugl-Meyer Upper Extremity (FM-UE) | Baseline, Change from Baseline at 8th week
  FM-UE is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia. It is applied clinically and in research to determine disease severity, describe motor recovery, and to plan and assess treatment.
Mobility Test: Timed Up and Go (TUG) | Baseline, Change from Baseline at 8th week
  This test is a general physical performance test used to assess mobility, balance and locomotor performance in elderly people with balance disturbances. More specifically, it assesses the ability to perform sequential motor tasks relative to walking and turning. This test is rated on a scale of second measurement, considering less than 10 second as "normal function" and more than 30 seconds as "severely abnormal function".
Balance Test: Balance Berg Scale (BBS) | Baseline, Change from Baseline at 8th week
  This scale is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It does not include the assessment of gait. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function.
Health-related quality of life Questionnaire: Short Form 36 (SF36) v2 | Baseline, Change from Baseline at 8th week
  This questionnaire evaluate general health status in eight domains: physical function, role physical, bodily pain, general health, vitality, social function, role emotional and mental health; which are also reduced to Physical and Mental Component Summary scores. Values above or below 50 (the normative score from the general population) are interpreted as better or worse than the reference population, respectively.
Functional capacity: 6 Minute Walk Test | Baseline, Change from Baseline at 8th week
  - 6 Minutes Walk Test: The 6MWT is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity. The measurement is considered by meters, so the more meters the user is able to get, the more distance and "normal functioning" will register.

SECONDARY OUTCOMES:
Level of physical activity questionnaire | Baseline, Change from Baseline at 8th week
  The global level of physical activity will be evaluated through the Global Physical Activity Questionnaire (GPAC). This tool covers several components of physical activity, such as intensity, duration, and frequency, and it assesses three domains in which physical activity is performed (occupational physical activity, transport-related physical activity, and physical activity during discretionary or leisure time). It is advised that show cards be used when the GPAQ is administered. Show cards should be developed for each of the activity types covered by the GPAQ: vigorous and moderate activity at work, transport activity, vigorous and moderate activity during leisure time, as well as sitting.
Sociodemographics questionnaire | Baseline
  Date of birth, gender, injury time of evolution and physical activity habits.
Anthropometric data - Weight | Baseline
  Weight (in kilograms). Weight and height will be combined to report BMI in kg/m^2)
Anthropometric data - Height | Baseline
  Height (in meters). Weight and height will be combined to report BMI in kg/m^2)

CONTACTS AND LOCATIONS:
Locations (1):
- Second Part Foundation, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided